CLINICAL TRIAL: NCT00441077
Title: Using a Communication Intervention to Provide Information About Inherited Risk to Underserved Latino Communities
Brief Title: Interventions to Educate An Underserved Population About Inherited Disease Risks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 999907102; 07-HG-N102
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-25

CONDITIONS: Healthy Volunteers
Keywords: Genetics; Family History; Latino; Information Seeking; Lay Health Advisors; Cancer; Heart Disease; Diabetes; Information
MeSH Terms: conditions — Neoplasms; Heart Diseases; Diabetes Mellitus | interventions — Educational Status

INTERVENTIONS:
Behavioral: Education

SUMMARY:
This study will examine how to communicate with an underserved population about inherited disease risks. It will present information about inherited risk to a Latino population through either a lay health advisor (LHA) or through printed information. The LHA is a member of the Latino community who has received training in public speaking, group facilitation, and managing group dynamics and in family health history and genetics. Previous studies have shown that an LHA can effectively communicate health information to diverse audiences, but such interventions have not been studied in the context of inherited risk.

Spanish-speaking Latino men and women over the age of 18 in the Oakland, CA, and Washington, DC, areas who have basic Spanish reading and writing skills may be eligible for this study.

Participants are recruited to one of two groups. One group participates in group educational sessions with an LHA about inherited disease risks and family health history, and the other receives this information from a brochure.

Educational Sessions

Groups of 5 to 8 individuals complete a questionnaire and then participate in a 45-minute educational session on concepts related to genetics, family health history, lifestyle and environment. Participants engage in role-playing to practice discussing family health history with family members. The LHA teaches participants the skills needed to fill in family health history tool called My Family Health Portrait and answers questions. After the question and answer session, participants complete a second questionnaire.

Brochure-Only

Participants complete a questionnaire and then read a Spanish-language brochure produced by the U.S. Surgeon General's Office about the importance of knowing one's family history. They then complete a second questionnaire.

DETAILED DESCRIPTION:
How to effectively educate the public about inherited risk is an important communication issue now and will likely become even more important over the next decade. Little research has been conducted, however, to examine how to communicate about this topic with individuals from underserved populations. The planned study provides a unique and innovative opportunity to examine how to reach an underserved community and present information about inherited risk in an understandable and usable form by building upon an existing relationship between NHGRI and the National Council of La Raza (NCLR). NCLR has previously designed a culturally tailored lay health advisor (LHA) intervention designed to increase knowledge and awareness about inherited risk among Latinos and to motivate them to seek information about their family history. The primary objective of this study will be to examine the pathways by which the LHA communication intervention impacts information seeking outcome variables. We will examine the roles of possible mediating variables (i.e., perceived information need, conceptual knowledge, self-efficacy) and assess the effects of contextual variables (i.e., family and personal history of disease, genetic beliefs, acculturation, health care access, sociodemographic variables) on the outcomes. The second objective is to provide quantitative data on the effects of the intervention on information seeking outcome measures (i.e., discussing family history with family members and health care providers) by comparing the intervention to a brochure-only condition; these data can inform the planning of a large-scale randomized controlled intervention trial. A third objective is to examine predictors of intention to seek information about family history at baseline. A quasi-experimental design will be used; we will recruit 350 individuals to participate in the LHA intervention and 200 to a brochure-only comparison group. All participants will be Spanish-speaking healthy volunteers who are at least 18 years of age and have basic Spanish reading and writing skills. Participants will be recruited through community-based clinics in Oakland, CA and Washington, DC and will either participate in a LHA or be asked to read information about family history. They will complete brief, self-administered questionnaires in Spanish before and after participating in the intervention or reading the brochure. Because of the quasi-experimental design, multiple logistic regression models will be used in the analysis in order to control for covariates. Understanding how to effectively inform underserved communities about inherited risk is a research area of critical importance if genomics is to be used to benefit the public health.

ELIGIBILITY:
* INCLUSION CRITERIA:

All participants in this study will be healthy volunteers. Eligibility criteria for participation in the study are the following: (1) being at least 18 years of age; and (2) being able to speak Spanish and having basic Spanish reading and writing skills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550
Dates: Start 2007-02-19; Primary Completion 2007-12-12 (Actual); Study Completion 2007-12-12 (Actual)

PRIMARY OUTCOMES:
Intentions to seek information about family history.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - La Raza, Oakland, California
  - La Clinica del Pueblo, Washington D.C., District of Columbia

REFERENCES:
- [Background] Balcazar H, Alvarado M, Hollen ML, Gonzalez-Cruz Y, Pedregon V. Evaluation of Salud Para Su Corazon (Health for your Heart) -- National Council of La Raza Promotora Outreach Program. Prev Chronic Dis. 2005 Jul;2(3):A09. Epub 2005 Jun 15. PMID 15963311
- [Background] Catz DS, Green NS, Tobin JN, Lloyd-Puryear MA, Kyler P, Umemoto A, Cernoch J, Brown R, Wolman F. Attitudes about genetics in underserved, culturally diverse populations. Community Genet. 2005;8(3):161-72. doi: 10.1159/000086759. PMID 16113533
- [Background] Derose KP, Baker DW. Limited English proficiency and Latinos' use of physician services. Med Care Res Rev. 2000 Mar;57(1):76-91. doi: 10.1177/107755870005700105. PMID 10705703